CLINICAL TRIAL: NCT00543946
Title: Ascending Single Dose Study of The Safety, Tolerability, Pharmacokinetics, of GAP-134 Administered Intravenously as a 24-Hour Infusion to Healthy Japanese Male Subjects
Brief Title: Single Ascending Dose of GAP-134 as a 24-hour IV Infusion in Healthy Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 3205K2-1002
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — 1-(2-aminoacetyl)-4-benzamidopyrrolidine-2-carboxylic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Drug: GAP-134 — 24-Hour IV infusion, SAD

SUMMARY:
This is a study of GAP-134, an antiarrhythmic di-peptide. This study will provide an initial assessment of the safety, tolerability, and pharmacokinetics (PK) of GAP-134 after administration of ascending single intravenous (IV) doses to healthy Japanese male subjects.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the most commonly occurring sustained arrhythmia in clinical practice. AF is a serious disorder associated with an increased risk of stroke, morbidity and mortality, and the number of patients is estimated to double within the next 4 decades. The currently available antiarrhythmic drugs have limited efficacy and are associated with serious side effects of which potentially lethal ventricular proarrhythmias are one of the major concerns. Thus, there is a large unmet clinical need for efficacious and safe antiarrhythmic drugs for the treatment of AF.

The classical orientation of antiarrhythmic therapy has been to modulate cardiac ion channels (sodium, potassium or calcium) or the autonomic nervous system. However, numerous experimental and clinical studies have suggested that cardiac conduction slowing and impaired gap junction intercellular communication (GJIC) are important in the pathogenesis of cardiac arrhythmias, including AF. General conduction slowing or the presence of small islands of intra-atrial conduction block resulting from a decreased gap junction conductance, altered gap junction expression and heterogeneous spatial distribution of gap junctions may provide turning points for the multiple waves, and thereby promote re-entry of impulses. In recognition of this, several authors have proposed gap junction modulation as a potential new target in the treatment of AF. GAP-134 is an antiarrhythmic dipeptide that has demonstrated in vitro and in vivo efficacy in mouse and dog models of arrhythmia. GAP-134 has no apparent proarrhythmic activity or hemodynamic compromise and does not show any significant binding in a panel of >60 different receptors and ion channels. If determined to be safe and effective the indication sought for GAP-134 will be the prevention of post operative atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria

* Healthy Japanese men age 20-45.
* BMI within 17.6 to 26.4 kg/m2 and body weight greater than or equal to 45 kg.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking within 48 hours before study day 1 until the end of the inpatient confinement period.

Exclusion Criteria

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article (e.g., resection of liver, kidney, gallbladder, or gastrointestinal tract).
* Acute disease state.
* Any history of clinically important cardiac arrhythmias. Family history of long QT syndrome, Torsades de Pointes or unexpected cardiac death.
* Any clinically important deviation from normal limits in physical examination, vital signs, 12-lead electrocardiograms (ECGs), or clinical laboratory test results. Creatinine levels must be less than or equal to the upper limit of normal at screening.
* Demonstration of a positive orthostatic test at screening. The definition of a positive test is a greater than or equal to 20 mm Hg decrease in systolic blood pressure, greater than or equal to 10 mm Hg decrease in diastolic blood pressure, or a greater than or equal to 30 bpm increase in pulse rate, after standing for 3 minutes.
* Positive serologic findings for human immunodeficiency virus (HIV) antigen and antibodies, hepatitis B surface antigen (HbsAg), and/or hepatitis C virus (HCV) antibodies.
* Positive findings of urine drug screen.
* History of any clinically important drug allergy or adverse drug reaction (e.g., relapsing dermatitis, drug hypersensitivity, drug allergy, hypersensitivity to ingredient in the test articles or angioedemas)
* Use of any investigational drug within 90 days before study day 1 or prescription drug within 30 days before study day 1.
* Consumption of any caffeine-containing products.
* Consumption of grapefruit or grapefruit-containing products within 72 hours before study day 1 until the end of the inpatient confinement period.
* Use of any over-the-counter drugs, including herbal supplements (except for the occasional use of vitamins less than or equal to 100% of the recommended daily allowance), within 14 days before study day 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the safety and tolerability of ascending, single IV doses of GAP-134 as 24-hour continuous infusions and as a single bolus injection in healthy Japanese male subjects. | 6 months

SECONDARY OUTCOMES:
The secondary objective is to provide the initial PK profiles of ascending single IV doses (24 hour and 1-minute) of GAP-134 taken under fasting conditions in healthy Japanese male subjects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Shinagawa-Ku, Tokyo, Japan